CLINICAL TRIAL: NCT03373825
Title: Rapid Self-Testing to Prevent Fentanyl Overdose Among Young People Who Use Drugs
Acronym: RAPiDS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1612001662
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Accidental Overdose of Opiate
Keywords: overdose prevention; opioid overdose; risk behavior; harm reduction
MeSH Terms: conditions — Opiate Overdose; Risk-Taking; Harm Reduction

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either ARM1 or ARM2 depending on when they enrolled in the study.
Who Masked: Participant
Masking Description: Participants in ARM1 were only aware of the use of the "Take home rapid drug test" as a urine test. Participants in ARM2, while instructed to test their drug residue, were aware of the ability to use the "take home rapid drug test" as a urine test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): 50 participants will receive a kit containing 10 Rapid Response fentanyl test strips. We will ask participants to use the take-home rapid drug test to test their urine for presence or absence of fentanyl.
  Interventions: Behavioral: Take home rapid drug test
- Arm 2 (Experimental): 50 participants will receive a kit containing 10 Rapid Response fentanyl test strips. We will ask the participants to use the take-home rapid drug test to test the residue of their drug (ie. instruct them to test bags, cookers, spoons, etc.) for the presence or absence of fentanyl.
  Interventions: Behavioral: Take home rapid drug test

INTERVENTIONS:
Behavioral: Take home rapid drug test — The Rapid Response fentanyl test strips will be offered as take-home rapid drug tests to all participants to assess the willingness to use take-home rapid drug tests and the feasibility of using such an intervention at home. Arm 1 will be offered one method of using the take-home rapid drug test (urine testing). Arm 2 will be offered a second method of using the take-home rapid drug test (testing drug residue).
  Other Names: Rapid Response fentanyl test strips

SUMMARY:
The research team will enroll 100 young adults who use cocaine, heroin, inject drugs, or purchase prescription medications on the illicit market in a pilot study to be known as the Rhode Island Young Adult Prescription and Illicit Drug Study (RAPIDS). Participants will be trained to use a take-home home rapid drug test to test for the presence or absence of fentanyl in their drug supply. Half of the enrolled participants will be asked to test their urine for presence or absence of fentanyl, and the other half will be asked to test their drug residue for presence or absence of fentanyl. All participants will receive up to 15 take-home rapid drug tests for fentanyl. A follow-up survey will examine and compare utilization of the tests between the two groups. The study will be guided by the information-motivation-behavioral skills (IMB) model of engagement in health behaviors. The IMB model hypothesizes that if a person possesses the information, motivation, and behavioral skills to act, there is an increased likelihood that she/he will fulfill and maintain the desired behaviors (behaviors that will reduce accidental overdose).

DETAILED DESCRIPTION:
The research team will administer a brief survey to ascertain behavioral, psychosocial, and clinical factors that may be related to non-prescription fentanyl (NPF) exposure among young people who use illicit drugs. The researchers will also characterize knowledge of and perceptions towards drugs contaminated with NPF, as well as the potential diversion of prescription fentanyl formulations (e.g., transdermal patches). After the interviewer-administered survey has been completed, participants will provide urine samples to determine recent exposure to NPF and other illicit drugs.

The research team will assess the acceptability and feasibility of "take home rapid drug tests" to test for fentanyl exposure among 100 participants from the target population. After the enrollment and baseline survey, participants will be provided with rapid drug tests that detect the presence or absence of fentanyl in their drug supply. Half the participants will be asked to test their urine to see if they have been exposed to a fentanyl-contaminated drug. The other half will be asked to test the residue of the drug that they intend to use. Study participants will then be asked to return in 2 weeks for a brief follow-up survey that will assess whether they used the self-tests, whether the technology was acceptable and easy to use, and whether and how a positive test result altered their drug-using and overdose prevention behaviors.

ELIGIBILITY:
Inclusion Criteria

* 18-35 years of age
* resident of Rhode Island
* able to complete interviews in English
* self-reported heroin, cocaine, injection drug use, or counterfeit prescription pill use in the past 30 days

Exclusion Criteria

-participants who exclusively misuse medications obtained from a physician or diversion from someone else's prescription

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Willingness to use the take-home rapid drug test | At 2 week follow-up
  Self-reported measure of willingness to use take-home rapid drug tests (compare Arm1 and Arm2), measured by response to Likert-scale survey question (Strongly Agree--Strongly Disagree).

SECONDARY OUTCOMES:
Current overdose prevention behaviors | At baseline enrollment
  Self-reported steps taken to avoid accidental overdose, measured by a "check all that apply" survey question (what they do to avoid an accidental overdose).
Number of take-home rapid drug tests conducted | At 2 week follow-up
  Self-reported number of take home rapid drug tests used by participant (Arm1 vs Arm2).
Change in overdose prevention behaviors | At 2 week follow-up
  Self-reported actions taken in response to the take home rapid drug test results, measured by a "check all that apply" survey question (what they did after they found out the drugs were laced with fentanyl).
Recent non-prescription fentanyl exposure | At baseline enrollment
  Self-reported from personal experience (belief that they had ever been exposed to fentanyl), measured by Likert-Scale survey question (Strongly Agree--Strongly Disagree).
Recent non-prescription fentanyl exposure | At 2 week follow-up.
  Self-reported measure from take home rapid drug test results (any positive result).
Prevalence of take home drug tests reporting the presence of fentanyl exposure | At 2 week follow-up
  Self-reported measure of the number of times they received a positive rapid drug test result.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon DL Marshall, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amlani A, McKee G, Khamis N, Raghukumar G, Tsang E, Buxton JA. Why the FUSS (Fentanyl Urine Screen Study)? A cross-sectional survey to characterize an emerging threat to people who use drugs in British Columbia, Canada. Harm Reduct J. 2015 Nov 14;12:54. doi: 10.1186/s12954-015-0088-4. PMID 26577516
- [Background] BTNX Inc. Rapid Reponse™ Multi-Drug Integrated Split Specimen Cup. 2016 [cited 2016 Sept 18]; Available from: http://www.btnx.com/Product.aspx?id=18240
- [Derived] Goldman JE, Waye KM, Periera KA, Krieger MS, Yedinak JL, Marshall BDL. Perspectives on rapid fentanyl test strips as a harm reduction practice among young adults who use drugs: a qualitative study. Harm Reduct J. 2019 Jan 8;16(1):3. doi: 10.1186/s12954-018-0276-0. PMID 30621699